CLINICAL TRIAL: NCT06087328
Title: Comparing the Effects of Augmented Doses of Nicotine Replacement Therapy on Quitting Cigarettes and E-cigarettes
Brief Title: CAN-DOSE Study: Cessation With Augmented Nicotine for Dual Use Of Smoking and E-cigarettes
Acronym: CAN-DOSE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00130184; IRG-19-137-20 (Other Grant/Funding Number: American Cancer Society Institutional Research Grant)
Record Dates: First submitted 2023-10-12; First posted 2023-10-17 (Actual); Results first posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Smoking Cessation; Electronic Cigarette Use; Cigarette Smoking
MeSH Terms: conditions — Smoking Cessation; Vaping; Cigarette Smoking

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A (Active Comparator): 21mg patch, qd + 4mg lozenge prn [minimum of 5 & up to 20 per day]
  Interventions: Drug: Regular Nicotine patch and lozenge dose
- Arm B (Active Comparator): 21mg patch + 14mg patch qd + 4mg lozenge prn minimum of 5 & [up to 30 per day]
  Interventions: Drug: Augmented Nicotine patch and lozenge dose
- Arm C (Active Comparator): 2 x 21mg patches qd + 4mg lozenges prn [minimum of 5 & up to 40 per day]
  Interventions: Drug: Augmented Nicotine patch and lozenge dose

INTERVENTIONS:
Drug: Regular Nicotine patch and lozenge dose — 1mg patch, qd + 4mg lozenge prn [minimum of 5 & up to 20 per day]
  Arms: Arm A
Drug: Augmented Nicotine patch and lozenge dose — 21mg patch + 14mg patch qd + 4mg lozenge prn [minimum of 5 & up to 30 per day] OR 2 x 21mg patches qd + 4mg lozenges prn [minimum of 5 & up to 40 per day]
  Arms: Arm B; Arm C

SUMMARY:
Many people smoke cigarettes and use e-cigarettes, and have a hard time stopping. Nicotine replacement therapy medications, such as nicotine patches and lozenges, have been shown to help people quit e-cigarette use. The purpose of the present study is to see how well nicotine patches and lozenges help people quit both smoking and vaping, and to determine if higher doses of the medication work best.

DETAILED DESCRIPTION:
Tobacco use is a leading cause of cancer death and disability in the US, thus tobacco control remains an important public health priority. Alternative tobacco products have grown popular in the past decade, including electronic cigarettes (e-cigarettes; vaping). E-cigarettes were initially marketed as an alternative to or means for smoking cessation and became popular amongst those currently smoking. Recent estimates suggest that 54% of those who vape are currently smoking (i.e., dual use). Despite this, there is a lack of empirically tested interventions for dual use cessation among the general adult population. In a prior pilot study, investigators found preliminary evidence that a standard dose of nicotine replacement therapy (NRT; 21mg patch+4mg lozenge) was sufficient at helping exclusive e-cigarette users quit vaping. However, dual users (individuals who smoke cigarettes and use e-cigarettes) did not respond similarly. The proposed project aims to compare three doses of NRT (21mg patch+4mg lozenge; 21+14mg patch + 4mg lozenges; 21+21mg patch + 4mg lozenges) with a sample of dual users who wish to quit smoking and vaping use in order to understand more about how NRT can help dual users quit tobacco.

ELIGIBILITY:
Inclusion Criteria:

* Age 18yrs +
* Daily nicotine-containing e-cigarette user (25+ days per previous month)
* E-cigarette use 5+ times/day
* E-cigarette use > 1year
* Smoking >1 cigarette on 5-7 days per week
* Interest in quitting smoking and e-cigarette within the next month (>7 on 10-point scale)
* Willingness to use NRT
* Able to receive text messages/email
* Mailing address in South Carolina.

Exclusion Criteria:

* Medical conditions contraindicated to NRT use (including pregnancy, past month myocardial infarction, current cardiac arrhythmia, current angina, uncontrolled vascular disease, or medical conditions in which consumption of phenylalanine is contraindicated)
* Individuals reporting current use of other nicotine-containing products and/or smoking cessation medications
* Those who vape non-nicotine substances
* Individuals unable to consent (e.g. significant cognitive deficit, non-English speaking).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2023-12-05 (Actual); Primary Completion 2024-11-05 (Actual); Study Completion 2024-11-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Palmer, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina - Charleston, Charleston, South Carolina, United States

REFERENCES:
- [Derived] Palmer AM, DeMass R, Rojewski AM, Bagley EM, Carpenter MJ, Smith TT, Toll BA. Augmented Doses of Nicotine Replacement Therapy: Feasibility for Dual Cigarette and E-Cigarette Cessation. Am J Prev Med. 2025 Aug;69(2):107664. doi: 10.1016/j.amepre.2025.107664. Epub 2025 May 21. PMID 40409566

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From December 2023-September 2024, 46 participants were recruited from online advertisements.
Pre-assignment Details: Following consent, all females underwent a pregnancy test to ensure final eligibility for the study prior to randomization.
Period: 28-Day Treatment
Arm/Group | Arm A | Arm B | Arm C
Started | 16 | 15 | 15
Completed | 9 | 12 | 11
Not Completed | 7 | 3 | 4
Not completed — Lost to Follow-up | 7 | 3 | 4
Period: 1-month Follow-up
Arm/Group | Arm A | Arm B | Arm C
Started | 9 | 12 | 11
Completed | 9 | 11 | 10
Not Completed | 0 | 1 | 1
Not completed — Lost to Follow-up | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A | Arm B | Arm C | Total
Number analyzed (Participants) | 16 | 15 | 15 | 46
Age, Continuous [Mean (Standard Deviation); unit: Years] | 38.1 (7.7) | 39.3 (11.8) | 36.0 (11.1) | 37.8 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 6 | 8 | 26
  Male | 4 | 9 | 7 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Participants self-reported ethnicity as Hispanic/Latino or Non-Hispanic/Latino. A 'Not Reported' category was included for missing responses.
  Participants
    Hispanic or Latino | 2 | 0 | 1 | 3
    Not Hispanic or Latino | 14 | 14 | 14 | 42
    Unknown or Not Reported | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants] — Participants self-reported race. Categories included: American Indian or Alaskan Native, Asian, Black or African American, White or Caucasian, and Multiracial. A 'Not Reported' category was included for completeness; Two participants did not provide race information and are included in the 'Not Reported' category.".
  Participants
    American Indian or Alaska Native | 0 | 0 | 0 | 0
    Asian | 0 | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
    Black or African American | 2 | 2 | 0 | 4
    White | 14 | 11 | 13 | 38
    More than one race | 0 | 1 | 1 | 2
    Unknown or Not Reported | 0 | 1 | 1 | 2
Dependence [Count of Participants; unit: Participants] — Dependence score was used as a stratification variable. Dependence Score was determined by the highest score between the Fagerstrom Test for Nicotine Dependence (FTND) or Roswell ENDS Nicotine Dependence Scale (eNDS) with "low" categorized as scores 1-5 and "high" categorized as 6-10, respectively.
  Participants
    Low | 2 | 2 | 2 | 6
    High | 14 | 13 | 13 | 40

OUTCOME MEASURES:

1. Primary Outcome: Days of Dual Use Abstinence
Description: Number of days participants self-report abstinence from both e-cigarettes and smoking.
Time Frame: Day 28, Day 56
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Arm A | Arm B | Arm C
Number analyzed (Participants) | 16 | 15 | 15
Days
  Dual Abstinence Days 1-28 | 3.8 (7.8) | 11.2 (8.7) | 6.9 (10.3)
  Dual Abstinence Days 1-56 | 4.6 (8.3) | 23.8 (20.9) | 16.1 (21.4)

2. Secondary Outcome: Reduction
Description: Calculate the reduction of e-cigarette use and smoking between groups from baseline to end of treatment.
Time Frame: Day 28, Day 56
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Arm A | Arm B | Arm C
Number analyzed (Participants) | 16 | 15 | 15
Days
  Reduction in Days of E-cigarette Use Before and During Treatment (Days 1-28) | 6.1 (10.5) | 13.5 (10.7) | 9.5 (11.0)
  Reduction in Days of Cigarette Use Before and During Treatment (Days 1-28) | 7.9 (13.2) | 16.4 (10.3) | 12.2 (12.9)
  Reduction in Days of E-Cigarette Use Before and After Treatment (Days 29-56) | 3.2 (8.6) | 12.5 (15.0) | 9.3 (13.6)
  Reduction in Cigarette Use Before and After Treatment (Days 29-56) | 8.2 (15.2) | 19.5 (13.0) | 12.4 (13.9)

3. Secondary Outcome: Safety (Adverse Events)
Description: Adverse events and outcomes between groups will be evaluated.
Time Frame: Day 28
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A | Arm B | Arm C
Number analyzed (Participants) | 16 | 15 | 15
Participants
  Any Adverse Event | 9 | 13 | 10
  Any Severe Adverse Event (self-reported severity rating) | 0 | 1 | 0
  Any Doctor/Clinic/Hospital Visit due to Adverse Event | 0 | 0 | 0

4. Secondary Outcome: Feasibility/Acceptability
Description: Feasibility and acceptability were assessed by the proportion of eligible participants who enrolled, and among enrolled participants, the proportion who completed the Day 28 survey and the proportion who completed ≥80% of daily surveys during treatment.
Time Frame: Day 28
Population: Participants in the 'Eligible and Contacted' arm were only assessed for enrollment; survey completion was not measured. Participants in the 'Enrolled' arm were only assessed for survey completion; enrollment was not measured. Therefore, some rows have zero analyzed counts because those measures were not applicable to that arm.
Measure: Count of Participants; unit: Participants
Groups:
- Eligible and Contacted: Participants who responded to the recruitment materials, completed the screening survey, and were determined eligible based on their responses.
- Enrolled: Participants who signed consent for the study and were randomized (and for females, met non-pregnancy criteria prior to randomization).
Arm/Group | Eligible and Contacted | Enrolled
Number analyzed (Participants) | 46 | 37
Participants
  Eligible & Contacted: number analyzed (Participants) | 46 | 0
  Eligible & Contacted: Enrolled | 46 | 0
  Eligible & Contacted: Completed Day 28 Survey | 0 | 0
  Eligible & Contacted: Completed >=80% of Daily Surveys | 0 | 0
  Enrolled: number analyzed (Participants) | 0 | 37
  Enrolled: Enrolled | 0 | 0
  Enrolled: Completed Day 28 Survey | 0 | 25
  Enrolled: Completed >=80% of Daily Surveys | 0 | 12

ADVERSE EVENTS:
Time Frame: Days 1-28 of the study (i.e., treatment period).
Description: Adverse events (i.e., NRT side effects) were captured via the SAFTEE (Systematic Assessment for Treatment Emergent Events) on daily surveys during treatment.
Arm/Group | Arm A | Arm B | Arm C
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 9/16 | 13/15 | 10/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (N=16) | Arm B (N=15) | Arm C (N=15)
Skin irritation (Skin and subcutaneous tissue disorders) | 1 | 2 | 2
Irritation of nose, throat, or eyes (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 3
Difficulty sleeping (Psychiatric disorders) | 3 | 6 | 2
Vivid dreams (Psychiatric disorders) | 4 | 7 | 3
Upset stomach (Gastrointestinal disorders) | 3 | 5 | 5
Dizziness (Nervous system disorders) | 2 | 4 | 2
Headaches (Nervous system disorders) | 6 | 7 | 2

LIMITATIONS AND CAVEATS:
Feasibility measures were assessed separately for two populations: eligible participants and enrolled participants. As a result, certain rows in the outcome table have zero analyzed counts because those measures were not applicable to that arm.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-10-03): https://cdn.clinicaltrials.gov/large-docs/28/NCT06087328/Prot_SAP_000.pdf
  • Informed Consent Form (2023-09-19): https://cdn.clinicaltrials.gov/large-docs/28/NCT06087328/ICF_001.pdf